CLINICAL TRIAL: NCT00546975
Title: Effect of Oral Nutritional Supplements With Specialized Nutrients on Functional Recovery and Morbidity After Gastrointestinal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Compliance unacceptably low.
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof Herbert Lochs, Charite University Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 07.33.CLI
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2007-10

CONDITIONS: Patients Following Gastrointestinal Surgery
Keywords: gastrointestinal surgery; nutritional intervention; functional status; quality of life

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Resource Support® Novartis
  Interventions: Dietary Supplement: Resource Support®
- 2 (Active Comparator): Resource Protein®, Novartis
  Interventions: Dietary Supplement: Resource Protein®
- 3 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resource Support®
  Arms: 1
Dietary Supplement: Resource Protein®
  Arms: 2
Dietary Supplement: Placebo
  Arms: 3

SUMMARY:
Nutritional supplementation in postoperative recovery is still debated. Functional impairment is known to develop both secondary to inflammatory processes or secondary to reduced nutritional intake (e.g. disease induced anorexia). Since major surgery represents a traumatic event, surgical patients are at increased risk of malnutrition due to starvation, activation of neuroendocrine stress axis, inflammation and the subsequent increase in metabolic rate. Gastrointestinal surgery in particular can create additional problems as it often directly affects and limits dietary intake postoperatively and these effects frequently continue after discharge. Whereas manifest malnutrition occurs in about 15% of general surgical patients and in about 40% of oncology patients, postoperative weight loss of 5 to 9% occur in all surgical patients during the first two months. Moreover studies have shown that the nutritional status generally declines in hospital and both functional and nutritional status deteriorate for two months after discharge in malnourished surgical patients.

Most studies that have investigated nutritional support in the surgical setting have concentrated on perioperative or short term postoperative supplementation and focussed on in-hospital infection and complication rate.

Hypothesis I:

Nutritional intake is decreased after surgery which results in an impaired nutritional status which in turn is associated with a decreased functional status. Protein rich nutritional supplementation is able to reverse nutritional depletion and restore functionality.

Hypothesis II:

Surgical stress leads to inflammation; inflammation - in addition to reduced nutritional intake - impairs functional status and increases morbidity. Anti-inflammatory, protein rich nutritional supplementation aims to prevent inflammatory complications and therefore improves functional status and reduces morbidity. In patients with high risk for inflammation, a higher effect of anti-inflammatory oral nutrition on recovery of functional status is expected.

This study aims to determine whether 4 week oral nutritional supplementation and/ or specialized nutrients is effective in restoring functional status and reducing morbidity in surgical patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are > 50 years of age and < 80 years
2. Patients who have signed a written Informed Consent (Appendix I) prior to admission to the study.
3. Patients who have an ECOG performance status (presurgery) of 0, 1 or 2 (Appendix II).
4. Patients able to orally consume 500 mL or more of liquid a day after adaption
5. Patients undergoing elective gastrointestinal surgery [e.g. Colorectal surgery: colectomy, hemicolectomy, proctectomy; Small bowel resection/surgery; liver resection, splenectomy, non-whipple pancreatic surgery]

Exclusion Criteria:

1. Patients who are > 80 years of age and < 50 years
2. Patients who have co-morbid conditions, uncontrolled metabolic conditions or psychiatric conditions that might make tolerance or evaluation of the feeding formula difficult;
3. Patients undergoing Whipple´s procedure, gastrectomy, oesophageal resection
4. Patients who get preoperative nutritional support
5. Patients taking supplements (EPA, DHA)
6. Any concomitant severe disease e.g.

   * Patients with respiratory failure (FEV<0.8l/sec)
   * Patients with renal failure (Cr > 3mg/dl or dialysis patients)
   * Patients with hepatic dysfunction (Child >A)
   * Patients with cardiac failure (NYHA > III)
7. Patients suffering from an intestinal obstruction or ileus
8. Patients with an Hb level of >8 g/dL experiencing gastrointestinal haemorrhaging
9. Patients with HIV
10. Patients requiring immunosuppression treatments
11. Pregnancy
12. Patients undergoing emergency surgery
13. Other patients determined by a study investigator to be inappropriate for enrolment in this study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Physical Component Summary (from SF 36 Quality of life questionnaire) | 4 weeks

SECONDARY OUTCOMES:
hand grip strength | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Lochs, MD, Principal Investigator — Charite Universitätsmedizin Berlin Dept. of Gastroenterology
Locations (1):
- Dept of Surgery CCM, Berlin, State of Berlin, Germany